CLINICAL TRIAL: NCT00104923
Title: Phase I Trial of Intravenous Fenretinide (4-HPR) for Patients With Hematologic Malignancies
Brief Title: Fenretinide in Treating Patients With Refractory or Relapsed Hematologic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: California Cancer Consortium (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000413887; P30CA033572 (NIH); CCC-PHI-42; NCI-6528; LAC-USC-0C-04-3; NCI-06-C-0227; NCI-P6820
Record Dates: First submitted 2005-03-03; First posted 2005-03-04 (Estimated); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Chronic Myeloproliferative Disorders; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm
Keywords: adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent small lymphocytic lymphoma; recurrent mantle cell lymphoma; Waldenstrom macroglobulinemia; adult grade III lymphomatoid granulomatosis; recurrent adult grade III lymphomatoid granulomatosis; secondary acute myeloid leukemia; recurrent adult Burkitt lymphoma; recurrent adult immunoblastic large cell lymphoma; refractory chronic lymphocytic leukemia; recurrent adult lymphoblastic lymphoma; recurrent adult Hodgkin lymphoma; refractory multiple myeloma; recurrent adult acute lymphoblastic leukemia; relapsing chronic myelogenous leukemia; chronic eosinophilic leukemia; primary myelofibrosis; chronic neutrophilic leukemia; essential thrombocythemia; polycythemia vera; stage II multiple myeloma; stage III multiple myeloma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; recurrent marginal zone lymphoma; splenic marginal zone lymphoma; recurrent adult acute myeloid leukemia
MeSH Terms: conditions — Myeloproliferative Disorders; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Congenital Abnormalities; Lymphoma, Follicular; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Mantle-Cell; Waldenstrom Macroglobulinemia; Burkitt Lymphoma; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Hodgkin Disease; Pdgfra-Associated Chronic Eosinophilic Leukemia; Primary Myelofibrosis; Leukemia, Neutrophilic, Chronic; Thrombocythemia, Essential; Polycythemia Vera; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, B-Cell, Marginal Zone; Leukemia, Myeloid, Acute | interventions — Fenretinide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: fenretinide — Current dose level as an IV continuous infusion via central line over 5 days. Cycle is repeated every 3 weeks for up to 6 cycles

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as fenretinide, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving fenretinide in a different way may kill more cancer cells.

PURPOSE: This phase I trial is studying the side effects and best dose of intravenous fenretinide in treating patients with refractory or relapsed hematologic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of intravenous emulsified fenretinide in patients with refractory or relapsed hematologic malignancies.
* Determine the toxic effects of this drug in these patients.
* Determine the pharmacokinetics and in vivo activity of this drug in these patients.
* Determine, preliminarily, disease or tumor response in patients treated with this drug.

OUTLINE: This is a pilot, dose-escalation, multicenter study.

Patients receive emulsified fenretinide IV continuously over 5 days. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients who achieve a complete or partial response may continue to receive fenretinide at the discretion of the study chair.

Cohorts of 1 patient receive accelerated escalating doses of fenretinide until 2 patients experience moderate toxicity (cumulative across all dose levels) OR 1 patient experiences dose-limiting toxicity (DLT). After completion of the accelerated dose-escalation portion, the standard dose-escalation portion begins. Cohorts of 3-6 patients receive escalating doses of fenretinide until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience DLT. At least 6 patients are treated at the MTD. An additional 12 patients are treated at the MTD.

After completion of study treatment, patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: Approximately 40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed diagnosis of 1 of the following hematologic malignancies:

  * Non-Hodgkin's lymphoma (NHL)
  * Hodgkin's lymphoma
  * Multiple myeloma
  * Acute lymphoblastic leukemia
  * Acute myeloid leukemia
  * Chronic hematologic malignancy with a poor prognosis (e.g., failed 3 prior standard therapies), including any of the following:

    * Chronic lymphocytic leukemia
    * Chronic myelogenous leukemia
    * Indolent NHL
    * Myeloproliferative disorders
* Refractory or relapsed disease, as defined by 1 of the following:

  * Resistant to standard therapy for refractory or relapsed disease
  * Progressed after standard therapy for advanced disease
* No effective treatment exists
* Measurable or evaluable disease
* No active CNS disease

  * Previously treated leptomeningeal disease or brain metastases allowed provided there is no evidence of remaining cancer by positron-emission tomography, MRI, or spinal fluid cytology

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* At least 3 months

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3 (unless due to bone marrow involvement of disease)
* Platelet count ≥ 75,000/mm^3 (unless due to bone marrow involvement of disease)
* Hemoglobin ≥ 8.0 g/dL (transfusion allowed)
* No coagulation disorders

Hepatic

* AST and ALT < 2.5 times upper limit of normal (ULN) (≤ 5 times ULN for patients with liver metastasis)
* Bilirubin ≤ 1.5 times ULN

Renal

* Creatinine ≤ 1.5 times ULN

Cardiovascular

* No major cardiovascular disease

Pulmonary

* No major respiratory disease

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective double-method contraception prior to study entry, during study, and for at least 6 months after study participation
* No uncontrolled systemic infection
* No uncontrolled hypertriglyceridemia (i.e., triglyceride level > 500 mg/dL)
* No known HIV positivity
* No known allergy to egg products
* No known familial hyperlipidemia disorders
* No previously undiscovered hypertriglyceridemia
* No poorly controlled diabetes

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* More than 2 weeks since prior chemotherapy except hydroxyurea

  * No concurrent hydroxyurea during study drug administration
* No other concurrent anticancer chemotherapy

Endocrine therapy

* No concurrent hormone-ablative agents
* No concurrent steroids
* No concurrent tamoxifen or any of its analogues

Radiotherapy

* No prior cranial radiotherapy
* More than 2 weeks since prior radiotherapy

Surgery

* More than 20 days since prior surgery except for biopsy

Other

* Recovered from all prior therapy
* More than 2 weeks since prior investigational agents
* No other concurrent investigational agents
* No other concurrent antineoplastic therapy
* No other concurrent antioxidants
* No concurrent herbal or other alternative therapies
* No concurrent vitamin supplements (e.g., vitamin A, ascorbic acid, or vitamin E)

  * Standard dose multivitamin allowed
* No other concurrent medications that may act as modulators of intracellular ceramide levels or ceramide cytotoxicity, sphingolipid transport, or p-glycoprotein or multidrug resistance protein 1 (MRP1) drug/lipid transporters, including any of the following:

  * Cyclosporine or any of its analogues
  * Verapamil
  * Ketoconazole
  * Chlorpromazine
  * Mifepristone
  * Indomethacin
  * Sulfinpyrazone
* No concurrent medications that may cause pseudotumor cerebri, including any of the following:

  * Tetracycline
  * Nalidixic acid
  * Nitrofurantoin
  * Phenytoin
  * Sulfonamides
  * Lithium
  * Amiodarone
* No concurrent medication to control hypertriglyceridemia

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2005-02; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose of fenretinide | participants will be followed for the duration of cycle 1, which is expected to be 3 weeks.
To describe the toxicities of fenretinide | participants will be followed for the duration of treatment, which is expected to be 18 weeks or less

CONTACTS AND LOCATIONS:
Overall Officials: Ann Mohrbacher, MD, Study Chair — University of Southern California
Locations (4):
- United States (4):
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Warren Grant Magnuson Clinical Center - NCI Clinical Trials Referral Office, Bethesda, Maryland
  - M. D. Anderson Cancer Center at University of Texas, Houston, Texas
  - Joe Arrington Cancer Research and Treatment Center, Lubbock, Texas